CLINICAL TRIAL: NCT05196217
Title: CAREGIVER KNOWLEDGE AND EXPERIENCE OF CHILDREN WITH CHEWING PROBLEMS
Brief Title: CAREGIVER KNOWLEDGE AND EXPERIENCE OF CHEWING PROBLEM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, Sena Nur Begen, MSc, Atılım University
Other Study IDs: GO 20/290-1
Record Dates: First submitted 2021-12-26; First posted 2022-01-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Caregiver Awareness; Chewing Problem
Keywords: caregiver; awareness; experience; chewing problem

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chewing is the process of making the food taken into the mouth as a bolus with rhythmic, coordinated, and sequential movements. To normal chewing function oral and perioral sensory integrity; adequate lip closure and intraoral pressure; intraoral bolus transport; normal structure and coordination of lips, palate, tongue, jaw joint, chewing muscles should be ensured. Problems that occur in bolus formation starting from taking food into the mouth are called chewing problems.

The underlying cause of the chewing problem can be very diverse. The chewing problem can be seen in genetic, neuromuscular, gastrointestinal pediatric diseases as well as cognitive, behavioral problems or in healthy children. Many different health professionals take part in the rehabilitation of the chewing problem, but the family is at the center of the rehabilitation. For this reason, the level of knowledge, experience, and approach of the family is very important.

The aim of this study is to determine the swallowing-chewing problem knowledge levels, experiences and approaches of the caregivers of the child with chewing problems.

ELIGIBILITY:
Inclusion Criteria:

* being a primary caregiver of oral feding children, followed about chewing and swallowing problem more than 6 months

Exclusion Criteria:

* Don't except participate to study

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Being a primary caregiver of oral feding children, followed about cheming and swallowimg problem more than 6 months.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
chewing awareness | 1 day
  A one-to-one interview will be held with the caregivers in a quiet room, accompanied by a voice recorder. During interview; caregivers perspective, experiences and knowledge of the child's chewing and swallowing problem will be ask. The interviews will continue for a minimum of 20 minutes until sufficient data is collected for thematic analysis. 15 participants will be included in the study.

SECONDARY OUTCOMES:
Chewing Function | 1 day
  Karaduman Chewing Performance Scale (KCPS) developed by developed by Arslan et al., chewing function is classified at 5 different levels between 0 - 4 (Level 0= normal chewing function, Level 4= The child cannot bite and chew).

CONTACTS AND LOCATIONS:
Overall Officials: Selen Serel Arslan, assoc. prof., Study Director — Hacettepe University Faculty of Physical Therapy and Rehabilitation Ankara, TURKEY; Sena N Begen, MSc, Principal Investigator — Atilim University, Facultyof Health Sciences Department of Physiotherapy and Rehabilitation

IPD SHARING:
Plan to Share IPD: No
For a qualitative content analysis, The thematic analysis process involved multiple distinct phases as described by Braun and Clarke: the stages of familiarizing yourself with your data, generating initial codes, searching for themes, reviewing themes, defining and naming themes, producing the report (1). First, all interviews will be transcribed. A researcher will check the manuscripts, correct ıf there any mistake and make them anonymous. After the codes are determined. 2 researchers will come together at weekly meetings to discuss and develop themes. This approach will continue until no new information becomes available (theoretical saturation).

REFERENCES:
- [Background] Serel Arslan S, Inal O, Demir N, Olmez MS, Karaduman AA. Chewing side preference is associated with hemispheric laterality in healthy adults. Somatosens Mot Res. 2017 Jun;34(2):92-95. doi: 10.1080/08990220.2017.1308923. Epub 2017 Apr 10. PMID 28393655
- [Background] Serel Arslan S, Aydin G, Alemdaroglu I, Tunca Yilmaz O, Karaduman AA. Reliability and validity of the Karaduman Chewing Performance Scale in paediatric neuromuscular diseases: A system for classification of chewing disorders. J Oral Rehabil. 2018 Jul;45(7):526-531. doi: 10.1111/joor.12642. Epub 2018 May 20. PMID 29727486
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative research in psychology. 2006;3(2):77-101.